CLINICAL TRIAL: NCT03070314
Title: Bioavailability of an Echinacea Product (Echinaforce® Junior) in Children With a Common Cold, Aged 4-12 Years After Intake of a Daily Dosage
Brief Title: Echinaforce Junior Bioavailability Trial
Status: Withdrawn | Phase: Phase 4 | Type: Interventional
Why Stopped: no participants could be recruited who were eager to donate blood for bioavailability despite prolongation of the study period.
Sponsor: A. Vogel AG (Industry)
Collaborators: University Children's Hospital, Zurich (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 5000121
Record Dates: First submitted 2017-02-22; First posted 2017-03-03 (Actual); Last update posted 2018-07-18 (Actual); Status verified 2018-07

CONDITIONS: Common Cold
Keywords: Echinacea; bioavailability; children
MeSH Terms: conditions — Common Cold

STUDY DESIGN:
Intervention Model Description: The study participants take 5 tablets Echinaforce junior at once one after another per os. registered in Switzerland for children from age of 4 -12 years Six capillary blood draws are taken at the following time points: Start (0), after 15, 30, 60, 90, 270 minutes and then analyzed on the amount of tetraen. Bioavailability parameters will thereafter be calculated.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Echinaforce junior (Experimental): Echinaforce is an ethanolic extract from Echinacea purpurea fresh plant and root. The product is registered in Switzerland for children from age 4 years on for Treatment and prevention of respiratory tract infections.
  Interventions: Drug: Echinaforce junior

INTERVENTIONS:
Drug: Echinaforce junior — Echinacea Purpurea Extract Pill, sweetened and with orange flavour

SUMMARY:
In this bioavailability trial should be shown that the one of the main active constituent in alcoholic echinacea extracts, the alkylamide dodeca-2E,4E,8Z,10E/Z-tetraenoic acid isobutylamide (short: tetraen) is bioavailable in children of different age groups after intake of 5 Echinaforce junior tablets.

DETAILED DESCRIPTION:
In this bioavailability trial should be shown that the one of the main active constituent in alcoholic echinacea extracts, the alkylamide dodeca-2E,4E,8Z,10E/Z-tetraenoic acid isobutylamide (short: tetraen) is bioavailable in children of different age groups after intake of 5 Echinaforce junior tablets.

Six capillary blood draws are taken at the following time points: Start (0), after 15, 30, 60, 90, 270 minutes and thereafter the bioavailability is measured and calculated.

ELIGIBILITY:
Inclusion Criteria:

* Children in the age group 4-12 years with an uncomplicated common cold (upper respiratory tract infection)
* First symptoms appeared within the last 72 hours
* Written consent given by the parents and verbal consent of children who are capable of judgement

Exclusion Criteria:

* Not able to fast 2 hours prior to the treatment
* intake of another preparation containing echinacea within the last 24 hours
* Participation in a clinical trial within the last 30 days
* any progressive systemic illness, including tuberculosis, leukemia, connective tissue diseases, multiple sclerosis, or other autoimmune diseases; or
* history of relevant allergy, including allergy to Compositae plants

Ages: 4 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 0 (Actual)
Dates: Start 2017-02-20 (Actual); Primary Completion 2018-06-30 (Actual); Study Completion 2018-06-30 (Actual)

PRIMARY OUTCOMES:
Peak Plasma Concentration (Cmax) | 270 minutes measurement
  Peak concentration of tetraen

SECONDARY OUTCOMES:
Area under the plasma concentration versus time curve (AUC) | 270 minutes measurement
  Area of tetraen in plasma versus time curve
Timepoint when Cmax is reached (tmax) | 270 minutes measurement
  timepoint when maximum tetraen concentration is reached

CONTACTS AND LOCATIONS:
Locations (1):
- University Children's Hospital (UZH-UCH), Infectiology, University of Zurich, Zurich, Switzerland

IPD SHARING:
Plan to Share IPD: No